CLINICAL TRIAL: NCT04966910
Title: Stay Connected: Testing an Intervention to Combat COVID-19 Related Social Isolation Among Seattle-area Older Adults
Brief Title: Stay Connected: Testing an Intervention to Combat Coronavirus-related Social Isolation Among Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael Pullmann, Research Associate Professor, Department of Psychiatry And Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00011051; 5P50MH115837-03 (NIH)
Record Dates: First submitted 2021-06-25; First posted 2021-07-19 (Actual); Results first posted 2023-12-14 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Depression; Anxiety; Loneliness
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stay Connected (Experimental): Menu-driven set of strategies to combat loneliness, anxiety and depression in older adults
  Interventions: Behavioral: Stay Connected
- Treatment as usual (Active Comparator): Treatment as usual in these practice settings typically includes regular check-in calls and offering resources and referrals
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Stay Connected — Stay Connected is a menu-driven set of strategies to combat loneliness, anxiety and depression in older adults based on behavioral activation principles.
  Arms: Stay Connected
Behavioral: Treatment as usual — Regular check-ins, resource/referral provision
  Arms: Treatment as usual

SUMMARY:
This study will use the University of Washington's ALACRITY Center's (UWAC) Discover, Design, Build, & Test (DDBT) method to develop and test an intervention to address the mental health health needs of older adults in senior housing ("clients") who are forced to not only shelter-in-place but cannot have family or other visitors during this time. Older people (those over 60 years in age) are especially vulnerable and are more likely to have severe - even deadly - coronavirus infection than other age groups. These facts led to the need to have older adults socially isolate in order to protect their health; visits with family and friends are limited, and in senior housing (independent, supported and assisted care residences) have limited such visits by family to one person a day. This necessary practice of social distancing, while addressing an important public health crisis, unintentionally creates social isolation and loneliness, another deadly epidemic amongst the older population. Even before COVID-19, social isolation and loneliness was a prominent mental health and social problem in the aged, one that is associated with increases in other chronic conditions, dementia and suicide. Effective interventions for social isolation exist but are difficult to access and may not address all the concerns older adults have about this particular period of social isolation. The purpose of this proposed study is to deploy an adaptation of Behavioral Activation Therapy called Stay Connected to treat depression in older adults. The adaptation will allow activity directors and staff ("clinicians") in these settings and senior centers to deliver the therapeutic elements of the intervention (behavioral activation) in the context of social distancing/shelter-in-place policies. Social workers in these settings will oversee the activity director and staff delivery of the intervention. The investigators are working with a variety of senior housing types (HUD certified and private systems) and senior centers in Skagit county (rural) and King county (urban) in Washington (WA) so that the resulting intervention is not tied to economic levels or access to digital technology.

DETAILED DESCRIPTION:
Clinicians and clients from 6 rural and urban senior communities or senior centers will participate in this study. Senior communities or senior centers will be randomized to receive training and materials in either Stay Connected or a resource guide. The investigators will work with 2 staff from each community or senior center and conduct baseline, 4 week and 9 week assessments with clinicians and 20 clients from each community setting (N=12 clinicians and 120 clients).

ELIGIBILITY:
Older Adult Participants

Inclusion Criteria:

1. 60 years of age or older
2. Physical and cognitive ability to complete interviews by phone or using video-chat technology (e.g., Zoom)
3. English speaking
4. Resident of participating Seattle-area senior living communities or member of Seattle-area senior centers
5. Ability to provide consent
6. Score of 5 or higher on Patient Health Questionnaire (PHQ-9) or score of 5 or higher on Generalized Anxiety Disorder Scale (GAD-7) or score of 6 or higher on University of California Los Angeles (UCLA) Loneliness Scale
7. No suicidal ideation

Exclusion Criteria:

1. Under the age of 60
2. Inability to physically and/or cognitively consent and/or participate in study procedures via phone, computer, and/or video call
3. Non-English speaking
4. Scores below inclusion cut-offs on PHQ-9, GAD-7, and UCLA Loneliness Scale

Staff Participants Inclusion Criteria

1. English-speaking
2. Staff members in administration, social work, and/or activities department in Seattle area senior living communities or senior centers
3. Physical ability to complete training in intervention and complete questionnaires by phone, computer, or video-chat technology

Exclusion Criteria

1. Non-English speaking
2. Unable to physically or cognitively consent and/or participate in study procedures via phone, computer, and/or video call (e.g., Zoom)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Arean, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Clinics, with one staff in each clinic
Groups:
- Stay Connected Clients: Menu-driven set of strategies to combat loneliness, anxiety and depression in older adults
  Stay Connected: Stay Connected is a menu-driven set of strategies to combat loneliness, anxiety and depression in older adults based on behavioral activation principles. This group is for the clients who received the intervention.
- Usual Care Clients: Treatment as usual in these practice settings typically includes regular check-in calls and offering resources and referrals
  Treatment as usual: Regular check-ins, resource/referral provision. This group is for the clients who received treatment as usual.
- Stay Connected Clinicians: Menu-driven set of strategies to combat loneliness, anxiety and depression in older adults
  Stay Connected: Stay Connected is a menu-driven set of strategies to combat loneliness, anxiety and depression in older adults based on behavioral activation principles. This group is for the clinicians who delivered the intervention.
- Usual Care Staff: Treatment as usual in these practice settings typically includes regular check-in calls and offering resources and referrals
  Treatment as usual: Regular check-ins, resource/referral provision. This group is for the clinicians who delivered treatment as usual.
Period: Baseline
Arm/Group | Stay Connected Clients | Usual Care Clients | Stay Connected Clinicians | Usual Care Staff
Started | 22; 2 Clinics, with one staff in each clinic | 18; 2 Clinics, with one staff in each clinic | 2; 2 Clinics, with one staff in each clinic | 2; 2 Clinics, with one staff in each clinic
Completed | 22; 2 Clinics, with one staff in each clinic | 18; 2 Clinics, with one staff in each clinic | 1; 1 Clinics, with one staff in each clinic | 2; 2 Clinics, with one staff in each clinic
Not Completed | 0; 0 Clinics, with one staff in each clinic | 0; 0 Clinics, with one staff in each clinic | 1; 1 Clinics, with one staff in each clinic | 0; 0 Clinics, with one staff in each clinic
Not completed — Participant did not complete measure | 0 | 0 | 1 | 0
Period: 4-Week Follow-Up
Arm/Group | Stay Connected Clients | Usual Care Clients | Stay Connected Clinicians | Usual Care Staff
Started (All enrolled participants at baseline were considered to start the 4-week follow-up time period.) | 22; 2 Clinics, with one staff in each clinic | 18; 2 Clinics, with one staff in each clinic | 0; 0 Clinics, with one staff in each clinic (Clinicians did not receive 4 week timepoint surveys) | 0; 0 Clinics, with one staff in each clinic (Clinicians did not receive 4 week timepoint surveys)
Completed | 17; 2 Clinics, with one staff in each clinic | 14; 2 Clinics, with one staff in each clinic | 0; 0 Clinics, with one staff in each clinic | 0; 0 Clinics, with one staff in each clinic
Not Completed | 5; 0 Clinics, with one staff in each clinic | 4; 0 Clinics, with one staff in each clinic | 0; 0 Clinics, with one staff in each clinic | 0; 0 Clinics, with one staff in each clinic
Not completed — Clients did not complete measure at this timepoint | 5 | 4 | 0 | 0
Period: 9-Week Follow-Up
Arm/Group | Stay Connected Clients | Usual Care Clients | Stay Connected Clinicians | Usual Care Staff
Started (All enrolled participants at baseline were considered to start the 9-week follow-up time period. Participants were not required to complete the 4-week follow-up to start and be considered for the 9-week follow-up.) | 22; 2 Clinics, with one staff in each clinic | 18; 2 Clinics, with one staff in each clinic | 2; 2 Clinics, with one staff in each clinic (Clinicians did not receive a 4 week survey, therefore the number of participants who started this period is not the same as the number who completed the previous period.) | 2; 2 Clinics, with one staff in each clinic (Clinicians did not receive a 4 week survey, therefore the number of participants who started this period is not the same as the number who completed the previous period.)
Completed | 19; 2 Clinics, with one staff in each clinic | 17; 2 Clinics, with one staff in each clinic | 2; 2 Clinics, with one staff in each clinic | 0; 0 Clinics, with one staff in each clinic
Not Completed | 3; 0 Clinics, with one staff in each clinic | 1; 0 Clinics, with one staff in each clinic | 0; 0 Clinics, with one staff in each clinic | 2; 2 Clinics, with one staff in each clinic
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Participant did not complete measure | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants contributing demographic data. While more participants provided outcome measures at baseline, several participants did not respond to the demographic questions at baseline.
Groups:
- Stay Connected Clients: Menu-driven set of strategies to combat loneliness, anxiety and depression in older adults
  Stay Connected: Stay Connected is a menu-driven set of strategies to combat loneliness, anxiety and depression in older adults based on behavioral activation principles.
- Usual Care Clients: Treatment as usual in these practice settings typically includes regular check-in calls and offering resources and referrals
  Treatment as usual: Regular check-ins, resource/referral provision
- Stay Connected Clinicians: Menu-driven set of strategies to combat loneliness, anxiety and depression in older adults
  Stay Connected: Stay Connected is a menu-driven set of strategies to combat loneliness, anxiety and depression in older adults based on behavioral activation principles. This group is the clinicians who delivered the Stay Connected intervention.
- Usual Care Clinicians: Treatment as usual in these practice settings typically includes regular check-in calls and offering resources and referrals
  Treatment as usual: Regular check-ins, resource/referral provision. this group is the clinicians who delivered usual care.
- Total: Total of all reporting groups
Arm/Group | Stay Connected Clients | Usual Care Clients | Stay Connected Clinicians | Usual Care Clinicians | Total
Number analyzed (Participants) | 17 | 14 | 1 | 2 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1 participant in the Usual Care arm did not contribute age data within the analytic sample.
  years
    number analyzed (Participants) | 17 | 13 | 1 | 2 | 33
    (all) | 74.4 (7.0) | 72.3 (4.9) | 28.0 | 38.0 (7.07) | 73.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Clinicians were not asked about their sex
  Participants
    number analyzed (Participants) | 17 | 14 | 0 | 0 | 31
    Female | 16 | 11 |  |  | 27
    Male | 1 | 3 |  |  | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 1 | 5
  Not Hispanic or Latino | 14 | 11 | 1 | 1 | 27
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 17 | 12 | 1 | 1 | 31
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Education Level [Count of Participants; unit: Participants]
  High school graduate or equivalent | 1 | 1 | 0 | 0 | 2
  Some college, no degree | 7 | 6 | 0 | 0 | 13
  Associate degree | 0 | 2 | 0 | 1 | 3
  Bachelors degree | 3 | 2 | 1 | 0 | 6
  Masters degree | 5 | 1 | 0 | 1 | 7
  Professional or doctorate | 1 | 2 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire (PHQ-9)
Description: The PHQ-9 consists of 9 depression items and one disability item. Each item is associated with a symptom of depression, which the participant rates whether or not they have experienced the symptom over the last two weeks, with severity rating of 0-3. It is one of the few measures that is brief (it takes less than one minute to give) and has been found to have excellent sensitivity to change over time. Older adult participants will complete this measure. Total score ranges from 0 - 27 and higher scores indicate higher levels of depression symptoms.
Time Frame: Baseline, 4-Week Follow-Up, and 9-Week Follow-Up
Population: Client participants contributing Baseline, 4-Week Follow-Up, and 9-Week Follow-Up data, excluding cases missing at any timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stay Connected Clients | Usual Care Clients
Number analyzed (Participants) | 17 | 14
score on a scale
  Baseline | 9.24 (6.08) | 7.29 (4.48)
  4-Week Follow-Up | 7.29 (4.55) | 6.29 (5.03)
  9-Week Follow-Up | 6.47 (5.08) | 7.50 (5.16)
Statistical Analysis 1: Comparison: Stay Connected Clients vs Usual Care Clients; Repeated measures ANOVA including a time x condition interaction term to test for differences in slopes by condition for client data; Test type: Superiority; p = 0.036, ANOVA — This p-value applies to the time x condition interaction variable in a repeated-measure ANOVA for client data

2. Primary Outcome: Generalized Anxiety Disorder (GAD-7)
Description: To assess for co-occurring anxiety, we will use the GAD-7, a 7- item screener for generalized anxiety. It consists of items related to GAD. Participants rate on a scale of 0-3 how much they have experienced in the last two weeks. The scale is a valid screener for GAD. Older adult participants will complete this measure. Total score ranges from 0 - 21, with higher scores mean an increased degree of severity of anxiety symptoms.
Time Frame: Baseline, 4-Week Follow-Up, and 9-Week Follow-Up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stay Connected Clients | Usual Care Clients
Number analyzed (Participants) | 17 | 14
score on a scale
  Baseline | 5.82 (5.64) | 4.43 (3.06)
  4-Week Follow-Up | 4.35 (4.11) | 3.71 (2.70)
  9-Week Follow-Up | 4.59 (5.10) | 4.93 (3.12)
Statistical Analysis 1: Comparison: Stay Connected Clients vs Usual Care Clients; Test type: Superiority; p = .226, ANOVA — This p-value refers to a time x condition interaction term in a repeated measures ANOVA

3. Primary Outcome: Sheehan Disability Scale (SDS)
Description: The SDS will be used as measure of disability/functional status. This is a brief analog disability scale, which uses visual-spatial, numeric and verbal anchors. The scale has been validated in medical and psychiatric populations with a variety of psychiatric diagnoses. Older adult participants will complete this measure. Total score ranges from 0 - 30, with higher scores indicating greater disruptions to their life from mental health symptoms.
Time Frame: Baseline, 4-Week Follow-Up and 9-Week Follow-Up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stay Connected Clients | Usual Care Clients
Number analyzed (Participants) | 17 | 14
score on a scale
  Baseline | 9.18 (9.36) | 8.29 (7.78)
  4-Week Follow-Up | 6.94 (8.72) | 7.21 (7.38)
  9-Week Follow-Up | 8.53 (9.45) | 9.71 (9.54)
Statistical Analysis 1: Comparison: Stay Connected Clients vs Usual Care Clients; Test type: Superiority; p = .674, ANOVA — This p-value refers to a time x condition interaction term in a repeated measures ANOVA to test for differences in slopes over time

4. Secondary Outcome: University of California Los Angeles (UCLA) Loneliness Scale
Description: A 3-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item as either O ("I often feel this way"), S ("I sometimes feel this way"), R ("I rarely feel this way"), N ("I never feel this way"). Older adult participants will complete this measure. Total scores range from 3 - 9, with higher scores indicating higher levels of loneliness.
Time Frame: Baseline, 4-Week Follow-Up, and 9-Week Follow-Up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stay Connected Clients | Usual Care Clients
Number analyzed (Participants) | 17 | 14
score on a scale
  Baseline | 6.53 (1.74) | 5.29 (1.27)
  4-Week Follow-Up | 5.53 (1.87) | 5.00 (2.00)
  9-Week Follow-Up | 5.88 (2.09) | 5.00 (1.66)
Statistical Analysis 1: Comparison: Stay Connected Clients vs Usual Care Clients; Test type: Superiority; p = .317, ANOVA — [p-value comment as in outcome 3, analysis 1]

5. Secondary Outcome: Behavioral Activation Scale (BADS)
Description: The Behavioral Activation for Depression Scale (BADS) can be used to track changes weekly in the behaviors hypothesized to underlie depression and specifically targeted for change by behavioral activation. It examines changes in the following areas: activation, avoidance/rumination, work/school impairment, and social impairment. The BADS consists of 25 questions, each rated on a seven-point scale ranging from 0 (not at all) to 6 (completely). Older adult participants will complete this measure. Total scores range from 0 - 150, with higher scores indicating more behavioral activation.
Time Frame: Client participants contributing Baseline, 4-Week Follow-Up, and 9-Week Follow-Up data, excluding cases missing at any timepoint.
Population: Participants contributing data at Baseline, 4-Week Follow-Up and 9-Week Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stay Connected Clients | Usual Care Clients
Number analyzed (Participants) | 17 | 14
score on a scale
  Baseline | 91.06 (26.25) | 94.64 (20.14)
  4-Week Follow-Up | 95.53 (25.01) | 99.01 (23.32)
  9-Week Follow-Up | 97.88 (18.58) | 97.71 (26.87)
Statistical Analysis 1: Comparison: Stay Connected Clients vs Usual Care Clients; Test type: Superiority; p = .741, ANOVA — [p-value comment as in outcome 3, analysis 1]

6. Secondary Outcome: Patient Reported Outcome Measurement Information System (PROMIS) Social Isolation - Short Version
Description: The PROMIS Social Isolation item bank assesses perceptions of being avoided, excluded, detached, disconnected from, or unknown by, others. This measure consists of 4 items, each rated on a five-point scale ranging from 1 - 5. Older adult participants will complete this measure. Total scores range from 4 - 20, with higher scores meaning more social isolation.
Time Frame: Baseline, 4-Week Follow-Up, and 9-Week Follow-Up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stay Connected Clients | Usual Care Clients
Number analyzed (Participants) | 17 | 14
score on a scale
  Baseline | 11.76 (3.82) | 10.50 (3.01)
  4-Week Follow-Up | 10.24 (3.31) | 9.71 (4.14)
  9-Week Follow-Up | 10.12 (3.60) | 9.43 (3.44)
Statistical Analysis 1: Comparison: Stay Connected Clients vs Usual Care Clients; Test type: Superiority; p = .737, ANOVA — [p-value comment as in outcome 3, analysis 1]

7. Secondary Outcome: Acceptability of Intervention Measure (AIM)
Description: This is a four item measure of intervention acceptability, where each item is rated on a 1-5 scale, with 1 = not at all acceptable and 5 = very acceptable, and the total score is a mean item score with minimum score of 1 and maximum of 5. Clinician participants complete this measure. Higher values are considered to be more positive (i.e., a more acceptable intervention).
Time Frame: Baseline and 9 week follow up
Population: Both Clinicians who delivered Usual Care dropped out of the study after baseline assessment. Only one clinician in the Stay Connected group completed baseline assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Stay Connected Clinicians: Clinicians who delivered a menu-driven set of strategies to combat loneliness, anxiety and depression in older adults
  Stay Connected: Stay Connected is a menu-driven set of strategies to combat loneliness, anxiety and depression in older adults based on behavioral activation principles.
- Usual Care Clinicians: Clinicians who delivered treatment as usual in these practice settings typically includes regular check-in calls and offering resources and referrals
  Treatment as usual: Regular check-ins, resource/referral provision
Arm/Group | Stay Connected Clinicians | Usual Care Clinicians
Number analyzed (Participants) | 2 | 2
score on a scale
  Baseline: number analyzed (Participants) | 1 | 2
  Baseline | 4.0 | 4.63 (0.53)
  9 week follow up: number analyzed (Participants) | 2 | 0
  9 week follow up | 4.38 (0.88) |

8. Secondary Outcome: Intervention Usability Scale (IUS)
Description: This is a ten item measure of how easy the intervention/system is to use and learn. Used for interventions (e.g., therapeutic modalities). Total scale scores range from 0 to 100, with higher scores considered to be more positive (i.e., a more usable intervention). Scores of 70 and higher are considered to be a usable intervention. Clinician participants complete this measure.
Time Frame: 9 weeks
Population: Data collected from Stay Connected group at 9 weeks only.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Stay Connected Clinicians: Menu-driven set of strategies to combat loneliness, anxiety and depression in older adults
  Stay Connected: Stay Connected is a menu-driven set of strategies to combat loneliness, anxiety and depression in older adults based on behavioral activation principles.
- Usual Care Clinicians: Treatment as usual in these practice settings typically includes regular check-in calls and offering resources and referrals
  Treatment as usual: Regular check-ins, resource/referral provision
Arm/Group | Stay Connected Clinicians | Usual Care Clinicians
Number analyzed (Participants) | 2 | 0
score on a scale | 85 (7.07) |

9. Secondary Outcome: Intervention Appropriateness Measure (IAM)
Description: This is a four item measure of how suitable an intervention is for the circumstances, where each item is rated on a 1-5 scale, with 1 = not at all appropriate and 5 = very appropriate, and the total score is a mean item score with minimum score of 1 and maximum of 5. Clinician participants complete this measure. Higher values are considered to be more positive (i.e., a more appropriate intervention).
Time Frame: Baseline, 9 week follow up
Population: Only clinicians were administered the measure. Both usual care clinicians dropped out of the study after baseline. Only 1 clinician in the Stay Connected group responded at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stay Connected Clinicians | Usual Care Clinicians
Number analyzed (Participants) | 2 | 2
score on a scale
  Baseline: number analyzed (Participants) | 1 | 2
  Baseline | 5.00 | 4.63 (0.53)
  9 weeks: number analyzed (Participants) | 2 | 0
  9 weeks | 5.00 (0) |

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the entirety of time patients were in the study from baseline to 9 week follow-up.
Groups:
- Stay Connected Clients: Clients receiving a menu-driven set of strategies to combat loneliness, anxiety and depression in older adults based on behavioral activation principles.
- Usual Care Clients: Clients receiving treatment as usual in these practice settings, typically including regular check-in calls and offering resources and referrals
- Stay Connected Clinicians: Clinicians delivering a menu-driven set of strategies to combat loneliness, anxiety and depression in older adults based on behavioral activation principles.
- Usual Care Clinicians: Clinicians delivering treatment as usual in these practice settings, typically including regular check-in calls and offering resources and referrals
Arm/Group | Stay Connected Clients | Usual Care Clients | Stay Connected Clinicians | Usual Care Clinicians
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/22 | 0/18 | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT04966910/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT04966910/SAP_001.pdf
  • Informed Consent Form (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT04966910/ICF_002.pdf